CLINICAL TRIAL: NCT04755491
Title: Chloride Transfer During Continuous Renal Replacement Therapy in the Intensive Care Unit: a Prospective Observational Cohort Study
Acronym: CLODICUS
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_1055
Record Dates: First submitted 2021-02-11; First posted 2021-02-16 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Acute Kidney Injury
Keywords: acute kidney injury; continuous renal replacement therapy; chloride transfer
MeSH Terms: conditions — Acute Kidney Injury | interventions — Continuous Renal Replacement Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Chloride transfer by continuous veno-venous hemofiltration: Chloride transfer over 24h of continuous veno-venous hemofiltration in mechanically ventilated ICU patients presenting with stage III AKI according to Kidney Disease: Improving Global Outcome (KDIGO) classification. Chloride concentrations will be measured in the serum, the urine, and the effluent of included patients every 4 to 6h from inclusion to H24.
  Interventions: Device: Continuous veno-venous hemofiltration
- Chloride transfer by continuous veno-venous hemodialysis: Chloride transfer over 24h of continuous veno-venous hemodialysis in mechanically ventilated ICU patients presenting with stage III AKI according to Kidney Disease: Improving Global Outcome (KDIGO) classification. Chloride concentrations will be measured in the serum, the urine, and the effluent of included patients every 4 to 6h from inclusion to H24.
  Interventions: Device: Continuous veno-venous hemodialysis
- Chloride transfer by continuous veno-venous hemodiafiltration: Chloride transfer over 24h of continuous veno-venous hemodiafiltration in mechanically ventilated ICU patients presenting with stage III AKI according to Kidney Disease: Improving Global Outcome (KDIGO) classification. Chloride concentrations will be measured in the serum, the urine, and the effluent of included patients every 4 to 6h from inclusion to H24.
  Interventions: Device: Continuous veno-venous hemodiafiltration

INTERVENTIONS:
Device: Continuous veno-venous hemofiltration — Treatment of KDIGO stage 3 AKI by CVVH, in which renal replacement therapy is applied using a convection technique (ultrafiltration). Indication, choice of CRRT modality, and CRRT settings are made by the clinician in charge, following international recommendations. The measurement of chloride transfer over 24h is performed during CVVH treatment.
  Groups: Chloride transfer by continuous veno-venous hemofiltration
Device: Continuous veno-venous hemodialysis — Treatment of KDIGO stage 3 AKI by CVVD, in which renal replacement therapy is applied using a diffusion technique (dialysis). Indication, choice of CRRT modality, and CRRT settings are made by the clinician in charge, following international recommendations. The measurement of chloride transfer over 24h is performed during CVVD treatment.
  Groups: Chloride transfer by continuous veno-venous hemodialysis
Device: Continuous veno-venous hemodiafiltration — Treatment of KDIGO stage 3 AKI by CVVHDF, in which renal replacement therapy is applied using a combination of diffusion technique (dialysis) and convection technique (ultrafiltration). Indication, choice of CRRT modality, and CRRT settings are made by the clinician in charge, following international recommendations. The measurement of chloride transfer over 24h is performed during CVVHDF treatment.
  Groups: Chloride transfer by continuous veno-venous hemodiafiltration

SUMMARY:
Acute kidney injury (AKI) is a frequently encountered complication in the intensive care unit (ICU), affecting on average 25 to 35% of patients. It is associated with an increased mortality, proportional to AKI severity. RRT induces important shifts of water and electrolytes. Thus, significant amount of chloride might unintentionally be transferred to patients.

Chloride is the main anion of the organism. It is involved in the regulation of numerous physiological processes. Thus, significant and rapid modification of chloride amount contained in the organism (as might be induced by renal replacement therapy) may be responsible for important, and potentially deleterious, consequences to critically ill patients.

Studies have shown that the administration of high amounts of chloride rich solutions (such as sodium chloride (NaCl) 0,9%) was associated with the development of hyperchloremic acidosis in a dose-dependent manner. This hyperchloremic acidosis could also be theoretically associated with deleterious physiological effects. However, the true clinical consequences of administration of high amounts of chloride rich solutions remains unclear. Their effect on mortality remains a matter of debate, the results of studies being very conflicting in that respect. Nevertheless, hyperchloremia itself and/or the rise of chloremia in the intensive care unit seems to be associated with increased mortality. Moreover, the impact of those chloride rich solutions on the development of acute kidney injury is also a subject of controversy, data from the literature being here again very conflicting.

A recent study already showed that continuous RRT (CRRT) techniques induce a significant transfer of sodium to patients benefiting from those techniques. In that study, the amount of sodium transferred depended mainly on the difference between patient's natremia and sodium concentration in dialysate and/or replacement fluid (usually higher than patient's natremia) used.

By analogy, it is likely that an occult transfer of chloride also happens during RRT, given the high chloride concentration of dialysate fluids (in continuous veno-venous dialysis, CVVD) and replacement fluids (in continuous veno-venous hemofiltration, CVVH), or when these 2 modalities are combined (continuous veno-venous hemodiafiltration, CVVHDF). Finally, the investigators suspect, although it remains undemonstrated so far, that the RRT technique (convective vs. diffusive) may influence this transfer, to an unknown extent. Nevertheless, this transfer and its potential determinants have never been studied yet.

If chloride overload (and its potential clinical consequences) induced by the administration of solutions such as NaCl 0,9% is being extensively studied, no study has ever focused on chloride transfer that may result from the use of renal replacement therapy. However, as mentioned above, it is very likely that such a chloride transfer to patients happens, and that its magnitude depends on different parameters such as RRT modality, RRT fluids characteristics, or patient's chloremia at the start of RRT.

The investigators conduct the present study to describe and compare the intensity of chloride transfer during the first 24 hours of renal replacement therapy by continuous veno-venous hemofiltration (CVVH), continuous veno-venous hemodialysis (CVVD),or continuous veno-venous hemodiafiltration (CVVHDF), and to determine if that transfer is more important with one or the other of those two techniques, in ICU patients affected with severe AKI requiring RRT. Secondary aims are to describe and compare the effects of chloride transfer under 3 RRT modalities (CVVD, CVVH and CVVHDF) on patient's outcome, organ failures, electrolyte and acid-base balance, fluid balance and hemodynamics. Finally, the investigators aim to develop a pharmacokinetic compartment model of chloride transfer during different modalities of RRT.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age > 18 years) affiliated to a social security regimen.
* Presenting with stage III AKI according to Kidney Disease: Improving Global Outcome (KDIGO) classification28.
* Treated with continuous RRT (CVVH or CVVD or CVVHDF) for less than 24 hours, whatever the method used.
* Mechanically ventilated at the time of inclusion in the study.

Exclusion Criteria:

* Patients on chronic hemodialysis / peritoneal dialysis.
* Patients on extracorporeal membrane oxygenation
* Patients on intermittent hemodialysis (acute or chronic)
* RRT initiated for a different reason than stage III AKI according to Kidney Disease: Improving Global Outcome (KDIGO) classification
* Withholding of life sustaining treatment concerning RRT, mechanical ventilation or cardiopulmonary resuscitation.
* Patients whose life expectancy is lower than 24 hours
* Patients under guardianship or another juridical protection
* Patient's or next of kin opposition to participate
* Patients previously included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will enroll all consecutive adult ICU patients, with stage III AKI (according to Kidney Disease: Improving Global Outcome (KDIGO) classification), and requiring continuous RRT (CVVH or CVVD or CVVHDF). Moreover, patients included will all be mechanically ventilated because of their initial clinical condition. This allows the selection of the most severe typology of ICU patients, in which the evaluation of chloride transfer may be the most relevant.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2022-08-24 (Actual); Study Completion 2022-08-24 (Actual)

PRIMARY OUTCOMES:
Amount of chloride (in mmol) transferred to the patient during the first 24 hours of RRT following inclusion | 24 hours after inclusion
  The amount of chloride transferred is defined as the difference between chloride input administered via the RRT generator (dialysate and CaCl2 in CVVD, or replacement fluid in CVVH, or both in CVVHDF), and the chloride mass eliminated in the form of effluent (ultrafiltrate or spent dialysate), aggregated throughout the first 24 hours following inclusion.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent BITKER, MD, PhD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital de la Croix-Rousse (Hospices Civils de Lyon) / Médecine Intensive - Réanimation, Lyon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chivot M, Bellomo R, Deniel G, Richard JC, Bitker L. Chloride Mass Transfers during Continuous Veno-Venous Hemodialysis with Regional Citrate Anticoagulation: Effects of Additional Ultrafiltration and Hamburger's Effect. Blood Purif. 2025;54(7):404-412. doi: 10.1159/000546322. Epub 2025 May 28. PMID 40435983